CLINICAL TRIAL: NCT00005952
Title: A Phase I/II Trial of Temodar in Pediatric Patients and Young Adults With High-Risk or Recurrent Solid Tumors
Brief Title: Temozolomide Plus Peripheral Stem Cell Transplantation in Treating Children With Newly Diagnosed Malignant Glioma or Recurrent CNS or Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1735; DUMC-1735-04-9R5; DUMC-1735-02-9R3; DUMC-1735-01-9R2; DUMC-1833-99-10; NCI-G00-1796; CDR0000067932 (Other: NCI)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Head and Neck Cancer; Kidney Cancer; Neuroblastoma; Ovarian Cancer; Sarcoma; Testicular Germ Cell Tumor
Keywords: childhood low-grade cerebral astrocytoma; recurrent childhood rhabdomyosarcoma; childhood craniopharyngioma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; stage IV Wilms tumor; stage V Wilms tumor; recurrent Wilms tumor and other childhood kidney tumors; childhood central nervous system germ cell tumor; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer; childhood germ cell tumor; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood choroid plexus tumor; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; untreated childhood supratentorial primitive neuroectodermal tumor; recurrent childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood medulloblastoma; recurrent childhood medulloblastoma; untreated childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway and hypothalamic glioma; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; newly diagnosed childhood ependymoma; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Testicular Germ Cell Tumor; Wilms Tumor; Testicular Neoplasms; Nasopharyngeal Neoplasms; Astrocytoma; Oligodendroglioma; Choroid Plexus Neoplasms; Medulloblastoma; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma | interventions — Filgrastim; Temozolomide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: temozolomide
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of temozolomide when given with peripheral stem cell transplantation and to see how well they work in treating children with newly diagnosed malignant glioma or recurrent CNS tumors or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of temozolomide in children with newly diagnosed malignant glioma or recurrent CNS or other solid tumors.
* Evaluate the toxicity of this treatment in these patients.
* Determine the activity of this treatment in these patients.

OUTLINE: This is a dose escalation study of temozolomide.

Patients receive filgrastim (G-CSF) subcutaneously (SQ) or IV beginning on day -5 and continuing through at least day 3. Peripheral blood stem cells (PBSC) are collected on days 0, 2, and 4. Patients then receive oral temozolomide daily for 5 consecutive days. PBSC collections are reinfused 1 day after the last dose of temozolomide. Patients also receive G-CSF beginning at the time of transplant and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicities.

Patients are followed every 3 months for 1-3 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed malignant glioma or recurrent malignant CNS tumor of any pathology OR
* Histologically confirmed non-CNS tumor

  * Recurrent soft tissue sarcomas (e.g., rhabdomyosarcoma)
  * Recurrent or resistant neuroblastoma
  * Recurrent Wilm's tumor
  * Recurrent Ewing's sarcoma
  * Recurrent primitive neuroectodermal tumors
  * Recurrent nasopharyngeal carcinoma
  * Recurrent germ cell tumor
* Expected cure rate less than 10% with standard therapy
* Measurable and/or active disease
* History of bone marrow tumor infiltration with or without mass lesions or isolated abnormal CSF cytology as only evidence of recurrent disease allowed if complete response was first achieved with primary conventional therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and under

Performance status:

* Karnofsky 70-100% OR
* Lansky 70-100%

Life expectancy:

* Greater than 8 weeks

Hematopoietic:

* Reasonably cellular bone marrow (greater than 15% cellularity on biopsy)
* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 75,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGPT less than 120 U/L

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* Systolic fraction or ejection fraction at least 80% predicted for age by echocardiogram

Pulmonary:

* CVC or DLCO at least 60% predicted for age OR clearance from pulmonologist

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active infection
* Able to tolerate vigorous hydration schedule

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent white blood cell transfusion
* No other concurrent hematopoietic growth factors

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No other concurrent cytotoxic drugs (systemic or intrathecal)

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 1 week since prior radiotherapy

Surgery:

* At least 1 week since prior surgery

Other:

* No other concurrent investigational agents

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2000-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Overall response at 12 months
Disease-free survival at 12 months

SECONDARY OUTCOMES:
Toxicity by NCI Common Toxicity Criteria v. 3.0 at 12 months
Engraftment related to autologous marrow or peripheral blood stem cell transplantation at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States